CLINICAL TRIAL: NCT00398567
Title: A Phase I/II Study of HKI-272 in Combination With Trastuzumab (Herceptin) in Subjects With Advanced Breast Cancer
Brief Title: A Phase 1/2 Study Of HKI-272 (Neratinib) in Combination With Trastuzumab (Herceptin) In Subjects With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-202 / B1891013
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Advanced Breast Cancer
Keywords: HKI-272; neratinib; trastuzumab; breast cancer; Nerlynx; PB-272; HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 - dose level 1 (160 mg) (Experimental): All subjects receiving HKI-272 dose level 1 in combination with trastuzumab
  Interventions: Drug: HKI-272; Drug: trastuzumab
- Part 1 - dose level 2 (240 mg) (Experimental): All subjects receiving HKI-272 dose level 2 in combination with trastuzumab
  Interventions: Drug: HKI-272; Drug: trastuzumab
- Part 2 - expanded MTD cohort (Experimental): All subjects receiving HKI-272 in combination with trastuzumab
  Interventions: Drug: HKI-272; Drug: trastuzumab

INTERVENTIONS:
Drug: HKI-272 — HKI-272 by mouth
  Other Names: neratinib
Drug: trastuzumab — trastuzumab 4 mg/kg IV as a loading dose followed by trastuzumab 2 mg/kg weekly thereafter
  Other Names: Herceptin

SUMMARY:
The purpose of this study is to determine the safety and efficacy of HKI-272 (neratinib) in combination with trastuzumab in patients with advanced breast cancer.

DETAILED DESCRIPTION:
Open label phase 1/2 study of ascending multiple oral doses of HKI-272 in combination with IV trastuzumab in subjects with advanced human epidermal growth factor receptor 2 positive (HER2+) breast cancer. Three to six subjects will be enrolled in each dose group. Adverse events and dose limiting toxicities will be assessed from the first dose of study drug though day 21. When the maximum tolerated dose (MTD) of HKI-272 plus trastuzumab is determined, an additional 30 subjects will be enrolled at that dose level, and followed for progression free survival for approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of breast cancer with current stage IIIB, IIIC or IV not curable by available therapy
* Progression following at least one Herceptin-containing cytotoxic chemotherapy regimen (neoadjuvant, adjuvant, or metastatic setting)
* HER2 positive breast cancer
* At least one measurable target lesion
* Adequate performance status
* Adequate cardiac, kidney, and liver function
* Adequate blood counts
* Willingness of all subjects who are not surgically sterile or post menopausal to use acceptable methods of birth control

Exclusion Criteria:

* More than 3 prior cytotoxic chemotherapy regimens for locally advanced or metastatic disease
* Major surgery, chemotherapy, radiotherapy, investigational agents, Herceptin or other cancer therapy within 2 weeks of treatment day 1
* Prior treatment with anthracyclines with cumulative dose of >400 mg/m^2
* Extensive visceral disease
* Active central nervous system metastases
* Pregnant or breast feeding women
* Significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom
* Prior exposure to HKI-272 or other HER2 targeted agents (except Herceptin and Tykerb)
* Significant cardiac disease or dysfunction
* History of life-threatening hypersensitivity to Herceptin
* Inability or unwillingness to swallow HKI-272 capsules
* Any other cancer within 5 years with the exception of contralateral breast cancer, adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-04-04 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2018-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (14):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - LAC/USC Medical Center, USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - City of Hope National Medical Center, Pasadena, California
  - University of Maryland, University of Maryland Medical Center, Baltimore, Maryland
  - Duke University, Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- China (5):
  - Chinese Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Tianjin Union Medicine Center, Tianjin, Tianjin Municipality
  - Cancer Hospital, Academy of Med Science and Peking Union Med, Beijing
  - 307 Hospital of Chinese People's Liberation Army, Beijing
  - Chinese PLA General Hospital, Beijing
- France (2):
  - Institut Curie, Paris
  - Centre Rene Gauducheau, Saint-Herblain
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib 160mg + Trastuzumab: All subjects receiving HKI-272 (neratinib) in combination with trastuzumab (Herceptin) HKI-272: neratinib 160 mg daily by mouth Herceptin: Herceptin 4 mg/kg IV as a loading dose followed by Herceptin 2 mg/kg weekly thereafter
- Neratinib 240mg + Trastuzumab: All subjects receiving HKI-272 (neratinib) in combination with trastuzumab (Herceptin) HKI-272: neratinib 240mg daily by mouth Herceptin: Herceptin 4 mg/kg IV as a loading dose followed by Herceptin 2 mg/kg weekly thereafter
- Part 2 - Expanded MTD Cohort: All subjects receiving HKI-272 (neratinib) in combination with trastuzumab (Herceptin) HKI-272: neratinib 240 mg daily by mouth Herceptin: Herceptin 4 mg/kg IV as a loading dose followed by Herceptin 2 mg/kg weekly thereafter
Period: Overall Study
Arm/Group | Neratinib 160mg + Trastuzumab | Neratinib 240mg + Trastuzumab | Part 2 - Expanded MTD Cohort
Started | 4 | 4 | 37
Completed | 0 | 0 | 3
Not Completed | 4 | 4 | 34
Not completed — Disease Progression | 3 | 4 | 27
Not completed — Withdrawal by Subject | 1 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Neratinib 160 mg + Trastuzumab; Neratinib 240 mg + Trastuzumab: All subjects receiving HKI-272 (neratinib) in combination with trastuzumab (Herceptin) HKI-272: neratinib 160 mg daily by mouth Herceptin: Herceptin 4 mg/kg IV as a loading dose followed by Herceptin 2 mg/kg weekly thereafter
- Total: Total of all reporting groups
Arm/Group | Neratinib 160 mg + Trastuzumab | Neratinib 240 mg + Trastuzumab | Part 2 - Expanded MTD Cohort | Total
Number analyzed (Participants) | 4 | 4 | 37 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.1) | 61.0 (12.8) | 50.5 (13.0) | 51.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 37 | 45
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 21 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 3 | 3 | 15 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: 16-week Progression-free Survival (PFS) Rate
Description: 16-week progression-free survival (PFS) rate for subjects with advanced breast cancer who receive neratinib at the maximum tolerated dose (MTD) in combination with trastuzumab, evaluable population.
Time Frame: From first dose date to progression status (PD or death) at 16-week
Population: The evaluable population was defined as the subjects who met the eligibility criteria for study enrollment, received at least 1 week of neratinib and at least 2 doses of trastuzumab, and had a baseline tumor assessment and at least 1 follow-up tumor assessment approximately 8 weeks after starting test article administration.
Measure: Number (95% Confidence Interval); unit: percentage of population
Arm/Group | Part 2 - Expanded MTD Cohort
Number analyzed (Participants) | 28
percentage of population | 44.8 [25.9 to 62.1]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Percentage of participants with partial response (PR) or complete response (CR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From first dose date to progression or last tumor assessment, up to five and a half years.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 - Expanded MTD Cohort
Number analyzed (Participants) | 28
percentage of participants | 28.6 [13.2 to 48.7]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was measured from the time at which response criteria were met for complete response (CR) or partial response (PR) (whichever status was recorded first) until the first date on which recurrence or PD was objectively documented, taking as the reference for PD the smallest measurements recorded since the test article administration started.
Time Frame: From start date of response to first PD, assessed up to five and half years after the first subject was randomized
Population: The subjects who had a complete response or partial response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 2 - Expanded MTD Cohort
Number analyzed (Participants) | 8
weeks | 44.2 [24.1 to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival was measured from the date of the first dose of test article until the first date on which recurrence or progression, or death due to any cause, was documented, censored at the last evaluation, investigator assessment.
Time Frame: From first dose date to progression or death, assessed up to five and half years.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 2 - Expanded MTD Cohort
Number analyzed (Participants) | 28
weeks | 15.9 [15.1 to 31.3]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The percentage of participants with a best overall response of a complete response (CR) or partial response (PR) or stable disease (SD) >=24 weeks.
Time Frame: From first dose date to progression or last tumor assessment, assessed up to five and half years.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 - Expanded MTD Cohort
Number analyzed (Participants) | 28
percentage of participants | 35.7 [18.6 to 55.9]

6. Secondary Outcome: Area Under the Curve of Neratinib Concentration
Description: Area Under the Curve of Neratinib concentration at day 22 following Administration of Neratinib 240 mg in combination with Trastuzumab 2 mg/kg in Subjects with Cancer.
Time Frame: Prior to the first dose, and at hours 1, 2, 4, 6, 8 and 24 on days 22.
Population: Subjects for whom complete blood samples at day 22 were available.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 2 - Expanded MTD Cohort
Number analyzed (Participants) | 33
ng*hr/mL | 1110 (430)

7. Secondary Outcome: Terminal-phase Elimination Half-life of Neratinib in Combination With Trastuzumab.
Description: Terminal-phase elimination half-life of Neratinib at day 22 following Administration of Neratinib 240 mg in combination with Trastuzumab 2 mg/kg to Subjects with Cancer.
Time Frame: Prior to the first dose, on days 22 through 23 of month 1, and on day 1 in months 2 through 6
Population: Subjects for whom complete blood samples at day 22 were available.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 2 - Expanded MTD Cohort
Number analyzed (Participants) | 27
hr | 21.22 (10.16)

ADVERSE EVENTS:
Time Frame: From first dose date through last dose date + 28 days.
Groups:
- Neratinib 240 mg + Trastuzumab; Part 2 - Expanded MTD Cohort: All subjects receiving HKI-272 (neratinib) in combination with trastuzumab (Herceptin) HKI-272: neratinib 240 mg daily by mouth Herceptin: Herceptin 4 mg/kg IV as a loading dose followed by Herceptin 2 mg/kg weekly thereafter
Arm/Group | Neratinib 160 mg + Trastuzumab | Neratinib 240 mg + Trastuzumab | Part 2 - Expanded MTD Cohort
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4 | 9/37
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 160 mg + Trastuzumab (N=4) | Neratinib 240 mg + Trastuzumab (N=4) | Part 2 - Expanded MTD Cohort (N=37)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 160 mg + Trastuzumab (N=4) | Neratinib 240 mg + Trastuzumab (N=4) | Part 2 - Expanded MTD Cohort (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 34
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 3 | 17
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 14
Asthenia (General disorders) | 0 | 0 | 13
Catheter site pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 1
Crying (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 6
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 1 | 0 | 4
Conjunctivitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 3
Haemoglobin decreased (Investigations) | 0 | 1 | 4
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 7
Weight increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 19
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 5
Dysgeusia (Nervous system disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 2 | 1 | 5
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3
Irritability (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 4
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 8
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less